CLINICAL TRIAL: NCT00914615
Title: Phase II Trial of Stereotactic Body Radiation Therapy for Unresectable Liver Metastases From Colorectal Carcinoma
Brief Title: Stereotactic Body Radiation Therapy (SBRT) in Liver Metastasis (COLD 3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 07-0348-C
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Liver Metastasis
Keywords: Stereotactic Body Radiation Therapy; Liver Metastasis from colorectal cancer; Patients with Liver Metastasis
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT for liver mets from colorectal cancer (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — Radiation therapy will be delivered on six occasions, over two weeks. Each treatment will take approximately 30 minutes to deliver (up to an hour including all imaging and set-up procedures). You may be asked to swallow 250 cc of oral contrast before each radiation therapy treatment. Pepto Bismol (a liquid that coats the stomach and is used to treat heartburn) and/or water may be combined with the contrast to improve the quality of the stomach's image.

SUMMARY:
This study is designed to see whether stereotactic body radiation therapy (SBRT) can reduce tumour size, slow progression of the disease, prolong life and improve quality of life. SBRT is concentrated focused radiation therapy delivered very precisely to the liver tumour.

Presently, the treatment for unresectable liver metastases from colorectal cancer is most often chemotherapy or novel targeted therapy. These treatments may improve survival, but not control the metastases permanently; so new treatments are needed to control metastases. It is hoped that knowledge obtained from this study will improve our ability to treat patients with liver tumours that cannot be treated with surgery and other methods, and that SBRT may prove to be a treatment that can lead to long-term and permanent control of liver tumours for some patients.

DETAILED DESCRIPTION:
From July 2003 to May 2007, over 50 patients with liver metastases participated in two studies at Princess Margaret Hospital (PMH) designed to determine the safety of treating liver metastases with SBRT. These studies have shown that SBRT can be delivered safely to the majority of patients with liver metastases. The treated tumour was controlled (shrank or remained the same size) in 74% of patients at one year following treatment. The median survival of patients was 16 months (i.e.half of patients survived longer and half shorter than 16 months). This survival rate is better than that expected in patients whose tumours grew bigger even though they were treated with chemotherapy. Supportive care only (no treatment other than care to make you feel better) in these patients is associated with a median survival rate of 6-12 months. We expect that the benefits of SBRT in this study will be similar to those observed in our initial studies.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have liver metastases from colorectal cancer 1) with histologic confirmation of metastases, 2) histologic confirmation of primary cancer and multiple new enhancing lesions in the liver consistent with metastases, or 3) histologic confirmation of primary cancer and a growing enhancing lesion in the liver Phase II SBRT Mets 13 consistent with a metastases
* Either 1) the tumour must be unresectable, based on the opinion of an experienced surgeon specializing in hepatic resection, or 2) the patient must be medically inoperable, or 3) extra-hepatic metastases must be present (making hepatic surgery an inappropriate treatment option).
* Karnofsky performance status (KPS) > 60 (Appendix II)
* Age: 18 years or older. Both male & female patients of all races can be included in this study. Female patients within reproductive years may not be, nor become, pregnant during participation in this study
* Patients must have recovered from the effects of previous therapy
* Maximal tumor size of 15 cm
* Adequate organ function as assessed as follows:

  * Hemoglobin > 90 g/L
  * Absolute neutrophil count > 1.0 bil/L
  * Platelets > 60bil/L
  * Bilirubin < 4.0 times upper range of normal
* INR < 1.5 or correctable with vitamin K (unless patients are on anticoagulation doses that have been stable for the past 2 months and they haven't had a bleed in the past 2 months)
* AST or ALT < 6.0 times upper limit of normal range
* Child's A 5-6 liver score
* Previous liver resection or ablative therapy is permitted
* Life expectancy > 3 months
* The volume of uninvolved must be at least 700 cc
* Up to five discrete liver tumors
* Patients must have signed a study-specific informed consent form. If the patient's mental status precludes this, written informed consent may be given by the patient's legal representative.

Exclusion Criteria:

* Patients with active hepatitis or encephalopathy related to liver failure
* Prior radiation therapy to the right upper abdomen, precluding reirradiation of the liver. That is, any previous radiation therapy in which a mean dose to the liver of 15 Gy in conventional fractionation was delivered, or previous doses to critical normal structures that would make re-irradiation unsafe. The PI should be called if there is any question of safety of re-irradiation.
* Prior uncontrolled, life threatening malignancy within the six months.
* Pregnancy is not permitted, and in women of child bearing age, a pregnancy test and acceptable methods of contraception are warranted.
* Previous variceal bleed within the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Determine one year local progression free rate, defined as lack of progression within the irradiated volume, using RECIST criteria. | 5 years

SECONDARY OUTCOMES:
Overall progression free survival | 5 years
Overall survival | 5 years
Quality of life | 5 years
CTC3.0 toxicity | 5 years
Cytokine response to radiation and association with complications | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada